CLINICAL TRIAL: NCT04040010
Title: The Effects of Bovine Colostrum in Bone Metabolism in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Petros Dinas (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor-Investigator, Petros Dinas, Senior Researcher in human physiology, University of Thessaly
Organization: University of Thessaly (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3. Colostrum & bone
Record Dates: First submitted 2019-07-26; First posted 2019-07-31 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Osteopenia; Osteoporosis
Keywords: bone metabolism; Postmenopausal women; bone markers; bovine colostrum; DXA
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Postmenopausal women colostrum supplement (Experimental)
  Interventions: Dietary Supplement: Colostrum supplementation for bone loss
- Osteoporosis patients colostrum supplement (Experimental)
  Interventions: Dietary Supplement: Colostrum supplementation for bone loss
- Osteopenia patients colostrum supplement (Experimental)
  Interventions: Dietary Supplement: Colostrum supplementation for bone loss
- Postmenopausal women placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Colostrum supplementation for bone loss
- Osteoporosis patients placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Colostrum supplementation for bone loss
- Osteopenia patients placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Colostrum supplementation for bone loss

INTERVENTIONS:
Dietary Supplement: Colostrum supplementation for bone loss — Participants in the interventions groups (i.e. colostrum supplementation) will take a colostrum mixture for 5 months (5 times per week; a total of 250ml per day in liquid form). Participants in the placebo groups (i.e. controls) will be taking a placebo mixture (a total of 250ml per day in liquid form per dose) for the same period of time.

SUMMARY:
Osteoporosis constitutes a major public health concern. For instance, in European Union 1 in 3 women and at least 1 in 6 men will suffer an osteoporotic fracture during their lifespan. The burden of osteoporosis is estimated to raise 25% by 2025. Worldwide, by 2050, the incidence of osteoporotic fractures is expected to increase 240% in women and 310% in men compared to 1990. The aforementioned estimates might indicate the existence of some gaps related to current products on the market for prevention and treatment of osteoporosis. Actually, the use of the approved pharmacological agents for osteoporosis have been decreasing in European Union and worldwide. Patients are becoming increasingly reluctant to take medicines; even those with severe osteoporosis are refusing treatment. Recent published reports on the matter revealed that patients fear the side effects of current pharmacological agents. Actually, therapy with bisphosphonates, the most prescribed medication for the treatment of postmenopausal, glucocorticoid-induced and male osteoporosis has been associated with severe side effects as osteonecrosis of the jaw and atypical femoral fractures.

Colostrum, a milky substance produced by mammals, known to be responsible for the development of the immune and skeleton systems of the offspring, has on its constituent's lactoferrin (LF). This multi-functional protein has been shown to affect both bone resorbing and bone formation pathways. The safety and tolerance on the use of bovine colostrum in humans (children and adults) have been well documented; it has a 'Generally Recognized As Safe' status from the United States Food and Drug Administration. Allergies and lactose intolerance, which are main shortcomings of milk consumption, have not been reported in relation to colostrum. Actually, human colostrum and bovine colostrum share the same bioactive components, but bovine sources are more potent than that of human. In accordance, bovine colostrum supplementation has been used in several therapeutic applications as gastrointestinal disorders, allergies and autoimmune diseases, viral and bacterial illnesses, and HIV-associated immunomodulation HIV. However, the effectiveness of bovine colostrum (as a whole and not only LF) to reduce bone losses has not been considered yet. Therefore, this study aims at analyzing the effects of bovine colostrum in diminishing bone mass losses in humans.

DETAILED DESCRIPTION:
Postmenopausal women (without any bone condition), osteopenia and osteoporosis patients (female and male) will be invited to join the study. Participants enrolling the project will be first measured on the following parameters: 1) general characteristics (age, sex, medical history); 2) bone mass parameters through Dual-energy X-ray absorptiometry (DXA); 3) bone formation and resorption markers (alkaline phosphatase, osteocalcin, N-telopeptides and urine deoxypyridinoline). After measuring the aforementioned parameters, consenting participants will be randomized into the following groups: Group 1: postmenopausal women taking colostrum supplementation; Group 2: postmenopausal women taking placebo; Group 3: osteopenia patients taking colostrum supplementation; Group 4: osteopenia patients taking placebo; Group 5: osteoporosis patients taking colostrum supplementation; Group 6: osteoporosis patients taking placebo. Power calculations (90% power, 0.05%) were performed in order to calculate the sample size needed in each group (considering stratification according to group, a minimum of 7 participants in each group are needed). Following 5 months intervention, participants will be re-assessed on the following parameters: 1) general characteristics (age, sex, medical history); 2) bone mass parameters through Dual-energy X-ray absorptiometry (DXA); 3) bone formation and resorption markers (alkaline phosphatase, osteocalcin, N-telopeptides and urine deoxypyridinoline).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (no menses for the last year at least);
* Osteoporosis patients (female): T-score<-2.5 at the femoral neck (or other anatomical site);
* Osteoporosis patients (male): T-score<-2.5 at the femoral neck (or other anatomical site)
* Osteopenia patients (female): T-score<-1.0 at the femoral neck (or other anatomical site);
* Osteopenia patients (male): T-score<-1.0 at the femoral neck (or other anatomical site)
* Patients taking drugs/ supplements for osteoporosis will be accepted in the study after going through a wash-up period

Exclusion Criteria:

* Women with irregular menses (i.e. with no established menopause)
* Patients taking medications for other diseases known to interfere with bone metabolism
* Patients with other chronic diseases (e.g. diabetes)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Change of alkaline phosphatase (μg/L) | Change from baseline of alkaline phosphatase at five months
  The alkaline phosphatase (μg/L) will be analyzed via human serum samples using an appropriate ELISA kit
Change of osteocalcin (μg/L) | Change from baseline of osteocalcin at five months
  The osteocalcin (μg/L) will be analyzed via human serum samples using an appropriate ELISA kit
Change of deoxypyridinoline (mmol/L) | Change from baseline of deoxypyridinoline at five months
  The deoxypyridinoline (mmol/L) will be analyzed via human serum samples using an appropriate ELISA kit
Change of C-terminal telopeptide (CTX) (pg/mL) | Change from baseline of C-terminal telopeptide at five months
  The C-terminal telopeptide (CTX) (pg/mL) will be analyzed via human serum samples using an appropriate ELISA kit
Change of bone mineral density (g/cm2) | Change from baseline of bone mineral density at five months
  The bone mineral density (g/cm2) will be analyzed via Dual-energy X-ray absorptiometry scan
Change of bone mineral content (gr) | Change from baseline of bone mineral content at five months
  The bone mineral content (gr) will be analyzed via Dual-energy X-ray absorptiometry scan

CONTACTS AND LOCATIONS:
Locations (1):
- FAME Lab, Department of Exercise Science, University of Thessaly, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Undecided